CLINICAL TRIAL: NCT03674723
Title: Application of the Indicator Amino Oxidation Technique for the Determination of Metabolic Availability of Methionine From Mung Beans, in Healthy Young and Older Adults
Brief Title: Metabolic Availability of Methionine From Mung Beans in Healthy Adults
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Glenda Courtney-Martin, Associate Scientist, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1000060319
Record Dates: First submitted 2018-09-14; First posted 2018-09-17 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Healthy
Keywords: Healthy; Men; Adults; Methionine
MeSH Terms: conditions — Multiple Endocrine Neoplasia Type 1 | interventions — Eating

STUDY DESIGN:
Intervention Model Description: Each subject will randomly receive 4 levels of methionine provided as free amino acids, Mung beans, or Mung beans combined with rice or wheat for a total of 10 studies x 3 days per study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Arms (Experimental): Methionine bioavailability in Mung beans Participants will be seen initially for pre-study assessment (3 hour). They will then be studied for up to 10 times. levels of phenylalanine intake (7 Study periods). You could be expected to participate in up to 10 different sets of experiments which will take 11 weeks to 6 months. Each set of experiment consists of a 3 day period. During the first 2 days (Adaptation Days) you will be expected to consume 4 meals per day consisting of a protein liquid drink and protein freecookies and/or a Mung bean stew with or without rice or wheat, which will be provided by the investigators
  Interventions: Other: Dietary Intakes

INTERVENTIONS:
Other: Dietary Intakes — Four levels of methionine intakes will be provided by the reference protein drinks, 3 levels of methionine from Mung beans and 3 levels from Mung beans with rice or wheat.

SUMMARY:
The research study is being done so we can determine the quality of the protein present in Mung beans. Amino acids are the building blocks of protein and protein quality is determined by the amount of amino acids present and by their bioavailability (their absorption and use by the body). Some amino acids are essential which means they must be obtained from the diet. If any one of the essential amino acids is missing in the diet, the body cannot make proteins that are used to repair tissue build bone, teeth, etc… Mung beans as a food source contain low amounts of the essential amino acid methionine which makes its protein incomplete. The amino acids in Mung beans are also affected by cooking. Our objective is to determine the amount of methionine in Mung beans that the body can use. We will test Mung beans by studying them after cooking them in a stew, on their own and by combining the Mung bean stew with rice or wheat in a mixed meal to make a more complete protein.

This research is being done in order to bridge the gap between knowledge of protein requirement and the amount of food needed to meet that requirement. Results from this study will be important for recommendations guiding food choices of Mung bean as a major protein source in the diet.

Previously the quality of dietary protein for human consumption was studied in animals. This study is being done in humans because studies in animals are not directly applicable to humans. Plant protein sources like Mung beans are important alternatives to animal protein in the diet. Plant protein consumption relative to animal protein can contribute to "enhance ecosystem resilience, and improved human health.

DETAILED DESCRIPTION:
If you agree to take part in this study, you will receive 3 different amounts of Mung beans which will contain different amounts of the essential amino acid methionine as well as 3 different amount of Mung beans complemented with rice or wheat. The Mung beans will be cooked in a stew served on its own or served with the rice or wheat. The quality of the protein in the Mung beans will be compared to the quality of a reference protein (egg protein) by giving you 4 reference diets containing amino acids patterned after the amino acid content of egg protein. The amount of Mung beans you receive will be provided in a random order.

Breath samples will be collected after the 4th meal in 15 min intervals for 1 hour. Breath collection will resume again two and a half hours after the 5th meal every 15 minutes until 30 minutes after the last meal. A total of 52 breath samples will be collected during each of the 3rd study day.

ELIGIBILITY:
Inclusion Criteria:

* Male, age 18 - 49 yrs, Healthy with no known clinical condition which would affect protein or AA metabolism, ex. Diabetes, Stable Body Weight (no more than 5 lb weight loss or gain in the past 3 months) Not on any medications that could affect protein or amino acid metabolism e.g. steroids

Exclusion Criteria:

* Unwillingness to participate or unable to tolerate the diet Recent history of weight loss within the last 3 months or on a weight reducing diet Inability to tolerate study diets (ex. Allergy to ingredients).

Ages: 18 Years to 49 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 6 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Metabolic availability of methionine in Mung beans | 2 years
  Apply the IAAO method to determine the MA of methionine in Mung beans prepared by moist cooking method.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Glenda Courtney-Martin, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No